CLINICAL TRIAL: NCT04104386
Title: The Impact of Personal Telomere Testing on Distress and Health Behaviors: A Randomized Controlled Trial of Women With Short and Average Telomere Lengths
Brief Title: Telomere Disclosure and Impact on Psychological Distress and Health Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Elissa Epel, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H11640-33841-01
Record Dates: First submitted 2019-06-19; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Telomere Length, Mean Leukocyte

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators were unfamiliar with who was categorized to which arm, and laboratory technicians were unfamiliar as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosure of Telomere Length Arm (Experimental): Telomere Length results were provided (personal value, means, and standard deviation of the group), and categorized as 'short' telomere length (bottom quartile) and 'not short' (above the bottom quartile) based on age related norms available from research literature.
  Interventions: Other: Telomere Disclosure Impact
- Non-Disclosure (No Intervention): Telomere Length results were not provided.

INTERVENTIONS:
Other: Telomere Disclosure Impact — Participants were either provided or not provided information about their personal telomere length and how they compared to the rest of the sample.
  Arms: Disclosure of Telomere Length Arm

SUMMARY:
There is now a critical mass of data linking health to telomere length, and blood telomere length is starting to become a commercially available measure, with several companies either offering or planning to offer this measure. With the growing intrigue and interest in telomeres and its commercial measurement, it is becoming increasingly important to understand the psychological and behavioral impact of receiving information about one's own telomere length. Therefore, the primary purpose of this study is to provide results of blood telomere length (from immune cells) to individuals, and to examine the subsequent psychological and lifestyle factors associated with learning one's personal results. Specifically, the investigators will assess if providing both telomere length and educational material on how cell aging is related to health and how it is modifiable, might lead to improvements in salutary health behaviors, and consequently, changes in telomere length.

A secondary goal of the study is methodological in nature. Human studies have mainly been limited to immune cells from blood, which requires a blood draw. The relation between blood telomere length and telomere length from other cells that are more easily accessible has not been assessed. Therefore, this study will assess relations between blood telomere length from venous blood draw with telomere lengths from buccal cells, hair follicle cells, and blood cells from a finger prick. This study will assess whether a new measure of telomere damage (TIFS) is related to other measures of cell aging. This study will also assess the reliability of the venous blood draw telomere length across three different assays (PCR, southern blot, and fluorescent in situ hybridization or FISH). To meet these aims, this study will collect samples of these cells from 240 healthy volunteers from the community.

DETAILED DESCRIPTION:
Background and Significance: Briefly sketch the scientific background leading to the present proposal, critically evaluate existing knowledge (with references), and specifically identify the gaps the project is intended to fill. State concisely the importance and health relevance of the research described in this application by relating the specific aims to the broad, long-term objectives.

Background and Rationale for Study:

There is now a comprehensive amount of data linking physical health to telomere length. Because of this, telomere length is becoming a commercially available measure. Several companies offer or plan to offer this measure; Spectracell Laboratories (www.spectracell.com) is one example of such a company. In order to have one's own telomere length measured, it's as easy as putting a zip code into a search function on their website to find the geographically closest clinician that will order the test. It is thus important to consider that there are no studies that have examined the possible responses to learning one's telomere length, whether it might be helpful or not, or even harmful. Learning about one's telomere length may motivate healthy behaviors, such as exercise or smoking cessation. The likely possibility of people learning their telomere length diagnostically in the future, and the potential for both positive and negative effects of learning this information, provide a strong rationale for studying the psychological and behavioral effects of learning one's telomere length.

Telomere length is a risk factor for disease:

Telomere length has become a valuable risk factor, as it is now linked to and predictive of many diseases and early mortality. For example, being of below average TL in a healthy population predicts threefold risk of earlier mortality in two studies. This effect size is comparable to other well accepted risk factors. Telomere shortening in these cases is likely acquired from lifetime exposures (lifestyle, cigarette smoking, infections) as well as from some presumably smaller genetic influence.

Telomeres can be very short from genetic/inherited conditions, and thus telomere testing can be helpful in the future to identify risk for rare genetically influenced conditions. Those with very short TL, probably in the bottom 5 to 10 percentile, are at risk of having a genetic defect in their genes that make telomerase (hTERT and hTR), and they may end up with haplosufficiency or half the normal dose of telomerase, which is not enough to protect telomeres from shortening. These defects are associated with short telomere syndromes, including liver fibrosis, lung fibrosis, bone marrow failure (aplastic anemia), poor immune function, and increased risk for cancers. Pulmonary Fibrosis (scarring of the lungs), a disease of aging which afflicts around 5 million people world wide, is characterized by short telomeres, and up to 15% of families with this condition have mutations in these genes for telomerase. Similarly, 3% of adults with aplastic anemia have telomerase mutations as well. If unrecognized and untreated, aplastic anemia quickly leads to death.

In sum, given the role of telomere shortening in common diseases, the evidence that healthy lifestyle behaviors are associated with longer telomere length, and the clear role of very short telomeres in rare conditions, telomere testing can potentially provide benefit to individuals.

Primary Aim 1: To assess whether learning one's personal blood telomere length (from immune cells) can have a positive impact on one's health behaviors and lifestyle factors (body weight, food choices, vitamin use, stress levels, and exercise). The investigators will further assess whether lifestyle and health behavior changes are related to subsequent changes in telomere length.

Telomere length has become commercially available and may become widely available in the coming years. Telomere length is a new biomarker that may or may not be helpful to know. It is related to lifestyle factors. The investigators have found high perceived stress is related to shorter TL, which several other labs have replicated, and the investigators now find that exercise buffers this relationship. Specifically, those high stress individuals who do vigorous exercise do not show shorter telomeres. Telomeres can also lengthen over time, as evidenced by recent evidence and the investigators unpublished data. A study found that improvements in lifestyle (including nutrition, stress reduction, and weight loss) were associated with increases in telomerase, the enzyme that lengthens telomeres. The investigators' unpublished data also shows that those who show decreases in stress over one year have increases in telomere length during this period, with a correlation of r = -.44. The investigators thus expect that improvements in lifestyle and stress levels can lengthen or at least forestall shortening of telomeres, and with a sample size of 240, the investigators can test these associations.

While the investigators are aiming to examine the behavioral and lifestyle effects of telomere length disclosure, of concern is whether receiving information about one's own blood telomere length could have a negative psychological impact. These concerns are quite valid, and a primary purpose of the present study, then, is to also examine the impact of finding out about one's blood telomere length on one's psychological well-being.

The investigators draw from a relevant study in the field of Alzheimers. In a 2009 study, investigators randomized 162 adult children of parents with Alzheimer's disease (thus at high risk of Alzheimers) to either a disclosure group, where they learned whether or not they tested positive for ApoE allele, a susceptibility risk factor for Alzheimer's Disease, and a nondisclosure group, where they did not learn of their results (The REVEAL trial). They measured anxiety, depression, and test anxiety at three points over the next year. Among those in the disclosure group, those who tested positive showed slightly greater test-related distress than the negative group, but the difference was not clinically meaningful. The findings support the psychological safety of disclosing genetic risk factor data, at least in this specific case.

More relevant to the investigators' current design was the REVEAL trial's primary outcome-- whether there were significant differences between the disclosure group and the nondisclosure group in distress. Importantly, there were no significant differences in measures of distress between the disclosure and nondisclosure groups. Further, those who discovered they were APOE-negative experienced psychological relief, showing lower test related distress compared to those who received no information about their APOE-negative status at 6 months. These results suggest that individuals who discover a genetic vulnerability to a disease are no more likely to experience psychological distress, and that those who are at no considerable risk actually experience relief, it is important to examine such processes related to a marker like telomere length which has been linked to a wide array diseases and disorders.

Learning about a risk factor like telomere length may or may not cause distress. The investigators' primary aim is to examine how being told one's own personal blood telomere length affects a person behaviorally and psychologically. The investigators expect it will cause only mild transient distress (slight increase on anxiety) if any, for those who are told they have short telomeres (bottom 25%). It is a susceptibility factor rather than a deterministic risk factor. In addition, learning about one's blood telomere length provides an opportunity for one to make behavior changes to improve blood telomere length, in contrast to a genetic risk factor that cannot change. Therefore, the investigators expect that people with short telomeres may be more motivated to increase healthy behaviors over the ensuing months. The investigators will emphasize that telomere length is changeable, and list the health behaviors that are associated with telomere length and thus may be linked to improvements in blood telomere length in a 'telomere information sheet.'

Behavior may change merely as a result of learning about the importance of telomeres and how they can take measures to protect their telomeres (in the "telomere information sheet"), regardless of knowing one's personal results. Therefore, it is necessary to have a control group for this educational portion of the study. Therefore, the investigators randomize one group to learn their telomere length only at the end of the study so that they can serve as a 'no result' control group for the study while the investigators assess behavior changes.

In addition to assessing emotional response when they are informed of their personal results, in the experimental group, the investigators will also assess whether the volunteers have made any changes in their health behaviors and lifestyle at either a 3 Month Follow-Up or 9 Month Follow-up from disclosure. The investigators will further examine, at 9 Month Follow-up, telomere length, by having participants return to the lab for a final blood draw. The investigators expect telomere length to change as a function of health behaviors and lifestyle changes that are undertaken and maintained throughout the 10 month period.

ELIGIBILITY:
Inclusion Criteria:

* 50-65 year old women

Exclusion Criteria:

* Women were excluded from the study if they had a major medical condition (cancer diagnosis in the past five years, cancer treatment within the past ten years, diagnosis of an autoimmune disorder) or reported currently smoking.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-04-04 (Actual); Primary Completion 2011-11-10 (Actual); Study Completion 2011-11-15 (Actual)

PRIMARY OUTCOMES:
Change sin Impact of Events Scale | 3 months
  Change in distress between groups in psychological distress between 1 week and 3 month followup. The IES scale quantifies the symptoms of distress into two sub-categories: Intrusion (7 items, max score 35) and Avoidance (8 items, max score 40). A subscale score ≥20 or a total score ≥40 indicates clinically significant levels of distress.

SECONDARY OUTCOMES:
change in health behaviors | 3 months post-randomization
  Composite Health Behaviors: At three time points (original blood draw, pre-randomization, and 3-month follow-up), we assessed (1) leisure time physical activity, (2) typical dietary practices, (3) sleep quality, and (4) mind-body activities. Since these measures exist on different scales, we harmonized the scores to be percentage of maximum possible. For example, a five-point scale was converted to (0%, 25% 50%, 75%, 100%), while a six-point scale was converted to (0%, 20%, 40%, 60%, 80%, 100%). This allowed us to meaningfully average scales using different Likert levels and create a mean composite score that weighed each component equally.
  (1) Leisure time physical activity was assessed with the leisure activity subsection of the Stanford Brief Activity Scale, a self-administered questionnaire developed for quick assessment of physical activity at work and during leisure activities over the past week,39 adjusted to past 3 months for the current study. Participants were provided five

IPD SHARING:
Plan to Share IPD: No